CLINICAL TRIAL: NCT04975945
Title: A Randomized Controlled Study Assessing Prolonged Parenteral Antibiotics Versus Single-time Intra-operative Intra-dermal Antibiotic Administration in Elective Clean and Clean-contaminated Surgeries for Prevention of Surgical Site Infections
Brief Title: Assessing Parenteral Antibiotics Versus Single-time Intra-operative Intra-dermal Antibiotic Administration for Prevention of SSI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Technical and organisational issues at the center, leading to inability to enrol study participants
Sponsor: The Grant Medical College & Sir J.J. Group of Hospitals (Other Government)
Responsible Party: Principal Investigator, Parth Bhavesh Gada, Junior Resident, The Grant Medical College & Sir J.J. Group of Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: generalsurgery/2021/01
Record Dates: First submitted 2021-07-21; First posted 2021-07-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2021-07

CONDITIONS: Surgical Wound Infection; Surgical Site Infection
Keywords: Ceftriaxone; Surgical wound infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local (Experimental): Participants will receive single-time intra-operative intra-dermal ceftriaxone (15-20mg/kg diluted in 10 ml normal saline)
  Interventions: Drug: Ceftriaxone Sodium
- Parenteral (Active Comparator): Participants will receive parenteral ceftriaxone (15-20mg/kg) for prolonged duration as per local protocol
  Interventions: Drug: Ceftriaxone Sodium

INTERVENTIONS:
Drug: Ceftriaxone Sodium — Intravenous vs local action

SUMMARY:
The purpose of the study is to study the incidence of surgical site infection when patients are given local versus parenteral antibiotics

DETAILED DESCRIPTION:
Patients undergoing above 18 years of age, giving consent and undergoing open or laparoscopic elective, CDC class I & II surgeries will be recruited. Cases will be randomised into two cohorts viz: parenteral antibiotic (Group A) vs single-time intra-operative intra-dermal antibiotic administration group (Group B). In operation theatre, after induction of anaesthesia, Group A will receive parenteral ceftriaxone (15-20mg/kg) whereas Group B will receive single-time intra-operative intra-dermal ceftriaxone (15-20mg/kg diluted in 10 ml normal saline). Post-operatively, incision site will be covered with occlusive dressing. First check-dressing will be done after 48 hours as per the existing institutional practices. After that surgical site will be inspected daily for wound infection. Patients with healthy wound will be discharged at the discretion of the treating surgeon and will be asked to follow up in General Surgery OPD weekly for one month. Cases who developed an SSI will have samples collected from the afflicted area for bacterial culture and antibiotic susceptibility testing. On development of SSI, the treating clinical team will commence antibiotic therapy as per their protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years
* Patients undergoing open and laparoscopic elective, CDC class I & II surgeries

Exclusion Criteria:

* Patients exhibiting hypersensitivity reaction to ceftriaxone
* Patients who are immunocompromised (retroviral disease and corticosteroid use)
* Patients not consenting to be a part of this study
* Pregnancy
* Febrile illness or leucocytosis at the time of surgery
* Planned for staged/multiple interventions during the hospital stay (endoscopies, image-guided biopsies etc)
* Patients with a possible septic focus distant from the surgical site such as diabetic foot ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical site infection | 1 month
  Infection occurs within 30 days after the operation and infection involves only skin or subcutaneous tissue of the incision and at least one of the following:
  1. Purulent drainage, with or without laboratory confirmation, from the superficial incision.
  2. Organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision.
  3. At least one of the following signs or symptoms of infection: pain or tenderness, localized swelling, redness, or heat and superficial incision is deliberately opened by surgeon, unless the incision is culture-negative.
  4. Diagnosis of superficial incisional SSI by the surgeon or attending physician
Organism isolated from wound | 1 month
  Microorganism grown on wound swab - Nominal data

SECONDARY OUTCOMES:
Total duration of hospital stay | 1 month
  Number of days of stay in the hospital - Ratio data (Numerical)

CONTACTS AND LOCATIONS:
Locations (1):
- Grant Government Medical College and Sir JJ Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
all IPD will be available after contacting the PI on parthg1895@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be available on completion of the study

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Akhter MS, Verma R, Madhukar KP, Vaishampayan AR, Unadkat PC. Incidence of surgical site infection in postoperative patients at a tertiary care centre in India. J Wound Care. 2016 Apr;25(4):210-2, 214-7. doi: 10.12968/jowc.2016.25.4.210. PMID 27064370
- [Background] Kotisso B, Aseffa A. Surgical wound infection in a teaching hospital in Ethiopia. East Afr Med J. 1998 Jul;75(7):402-5. PMID 9803631
- [Background] Young PY, Khadaroo RG. Surgical site infections. Surg Clin North Am. 2014 Dec;94(6):1245-64. doi: 10.1016/j.suc.2014.08.008. Epub 2014 Oct 3. PMID 25440122
- [Background] Holtz TH, Wenzel RP. Postdischarge surveillance for nosocomial wound infection: a brief review and commentary. Am J Infect Control. 1992 Aug;20(4):206-13. doi: 10.1016/s0196-6553(05)80148-8. PMID 1524269
- [Background] Patel IH, Kaplan SA. Pharmacokinetic profile of ceftriaxone in man. Am J Med. 1984 Oct 19;77(4C):17-25. PMID 6093513